CLINICAL TRIAL: NCT02404961
Title: Immunological Factors and Risk of Vulvodynia
Brief Title: Women's Health Study: Immunological Factors and Risk of Vulvodynia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0907M69161; 5R01HD058608 (NIH)
Record Dates: First submitted 2015-03-20; First posted 2015-04-01 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous Blood and Vulvar punch biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control (no vulvodynia): Clinically-confirmed as a woman with no history of vulvodynia.
  Interventions: Other: Vulvodynia
- Vulvodynia Case: Clinically-confirmed as a woman with vulvodynia.
  Interventions: Other: Vulvodynia

INTERVENTIONS:
Other: Vulvodynia — Comparison of reproductive, gynecological and environmental exposures, psychological trauma and psychiatric morbidity, and biological markers of immuno-inflammation and nerve fiber proliferation between cases and controls to determine potential etiology of vulvodynia.

SUMMARY:
The investigators plan to study the etiology of vulvodynia, a condition characterized by chronic vulvar discomfort, most often described as burning pain, occurring in the absence of relevant visible findings or a specific, clinically identifiable, neurologic disorder. Our hypothesis is that vulvodynia is the result of an altered immuno-inflammatory response mechanism that occurs as a consequence of reproductive, gynecologic, environmental, or psychological exposures, with abnormal vaginal microflora and genetic polymorphisms as potential modifiers of the effects of interest. Therefore, the investigators propose to collect information about reproductive, gynecological and environmental exposures, psychological trauma and psychiatric morbidity, and biological markers of immuno-inflammation and nerve fiber proliferation.

DETAILED DESCRIPTION:
Women aged 18-40 years who were seen for any reason within a 2-year period at one of the Twin Cities metro-area's Fairview Health Services outpatient clinics will be send a confidential self-administered questionnaire, and given the option to return it by mail, or complete it via phone or via a secure online server. This questionnaire will serve to determine any history of unexplained vulvar pain. Those with a history of past or current vulvar pain likely to represent vulvodynia, will be asked to come to one of four study clinic locations to confirm the diagnosis of vulvodynia. If confirmed, they will be asked to provide venous blood and vulvovaginal specimens. In addition, they will be asked to complete a medical history and psychosocial survey, along with an interviewer-administered Structured Clinical Interview for the Diagnostic and Statistical Manual-IV (SCID-IV). A random sample of women with no history of vulvar pain will be asked to serve as controls. Those confirmed as controls will also be asked to provide the same biological specimens and complete the same questionnaires/interview.

The long-term objective of this research is to provide etiological information that may prove critical to the treatment and prevention of vulvodynia, an under-recognized and extremely debilitating condition that we and others have shown may affect up to 10% of the adult female population.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed vulvodynia
* Women with no history of vulvar discomfort and clinically confirmed as acceptably control.

Exclusion Criteria:

* Women with vulvar pain attributed to a known cause.
* Women with any active gynecological yeast, bacterial, or viral infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18-40 years who were seen for any reason within a 2-year period at one of the metro-area's Fairview Health Services outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 30675 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reproductive, gynecological and environmental exposures and their association with vulvodynia & immuno-inflammatory response | Baseline
  Determine whether reproductive, gynecological and environmental exposures influence the odds of vulvodynia, and whether the effect is associated with immuno-inflammatory response
Past psychological trauma and psychiatric morbidity and their association with vulvodynia & immuno-inflammatory response | 6 month post baseline visit
  Determine whether psychological trauma and psychiatric morbidity influence the odds of vulvodynia and whether the effect is associated with immuno-inflammatory response
immuno-inflammation and nerve fiber proliferation and vulvodynia. | Baseline
  Determine whether markers of immuno-inflammation and nerve fiber proliferation are directly associated with the odds of vulvodynia, and, whether genetic and microbiological markers modify associations, as well as associations evaluated in aims 1 and 2 above.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Harlow, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Background] Nguyen RH, Turner RM, Rydell SA, Maclehose RF, Harlow BL. Perceived stereotyping and seeking care for chronic vulvar pain. Pain Med. 2013 Oct;14(10):1461-7. doi: 10.1111/pme.12151. Epub 2013 Jun 6. PMID 23742116
- [Background] Nguyen RH, Turner RM, Sieling J, Williams DA, Hodges JS, Harlow BL. Feasibility of collecting vulvar pain variability and its correlates using prospective collection with smartphones. Pain Res Treat. 2014;2014:659863. doi: 10.1155/2014/659863. Epub 2014 Jun 10. PMID 25006458
- [Result] Harlow BL, Kunitz CG, Nguyen RH, Rydell SA, Turner RM, MacLehose RF. Prevalence of symptoms consistent with a diagnosis of vulvodynia: population-based estimates from 2 geographic regions. Am J Obstet Gynecol. 2014 Jan;210(1):40.e1-8. doi: 10.1016/j.ajog.2013.09.033. Epub 2013 Sep 28. PMID 24080300
- [Result] Nguyen RH, Reese RL, Harlow BL. Differences in pain subtypes between Hispanic and non-Hispanic white women with chronic vulvar pain. J Womens Health (Larchmt). 2015 Feb;24(2):144-50. doi: 10.1089/jwh.2014.4892. Epub 2015 Jan 20. PMID 25603224